CLINICAL TRIAL: NCT06206720
Title: A Randomized, Double-blind, Placebo-controlled Phase II/III Clinical Trial to Evaluate the Safety and Efficacy of Deuremidevir Hydrobromide for Suspension in Hospitalized Infants Infected With Respiratory Syncytial Virus.
Brief Title: A Study of Deuremidevir Hydrobromide for Suspension in Chinese Infants Hospitalized With RSV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV116-RSV-II/III-01
Record Dates: First submitted 2023-12-28; First posted 2024-01-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Suspensions; GS-621763

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deuremidevir Hydrobromide for Suspension (Experimental): Deuremidevir Hydrobromide for Suspension will be orally administered at the dosing levels of 15 mg/kg BID, 20 mg/kg BID, or 20 mg/kg TID for five days according to the weight of patients.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension
- Placebo (Experimental): Placebo will be orally administered at the dosing levels of 15 mg/kg BID, 20 mg/kg BID, or 20 mg/kg TID for five days according to the weight of patients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide for Suspension — 15 mg/kg BID group: 15 subjects will receive Deuremidevir Hydrobromide for Suspension once every 12 hours, total 10 times.
  20 mg/kg BID group: 15 subjects will receive Deuremidevir Hydrobromide for Suspension once every 12 hours, total 10 times.
  20 mg/kg TID group: 15 subjects will receive Deuremidevir Hydrobromide for Suspension 3 times every day, total 15 times.
  Other Names: VV116
  Arms: Deuremidevir Hydrobromide for Suspension
Drug: Placebo — 15 mg/kg BID group: 5 subjects will receive placebo once every 12 hours, total 10 times.
  20 mg/kg BID group: 5 subjects will receive placebo once every 12 hours, total 10 times.
  20 mg/kg TID group: 5 subjects will receive placebo 3 times every day, total 15 times.
  Other Names: VV116 placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety, efficacy, pharmacokinetic (PK) characteristics and antiviral activity of different doses of Deuterium Hydrobromide for suspension in the treatment of respiratory syncytial virus infection in infants.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, placebo-controlled, dose-ascending trial, and the subjects are infants infected with RSV from 1 to 24 months.

It is estimated that 60 subjects will be included and divided into low-dose group (15 mg/kg，BID), middle-dose group (20 mg/kg,BID) and high-dose group (20 mg/kg,TID), with 20 cases in each group, and they will be randomly assigned to the experimental drug group and the placebo group according to the ratio of 3: 1.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female infants ≥1 month and ≤24 months；
2. Diagnosis of RSV infection by antigen detection or nucleic acid within 36 hours preceding initial dosing；
3. Onset of RSV infection symptoms should be ≤ 5 days；
4. Patient must weigh ≥ 2.5 kg and ≤ 20 kg at screening；
5. Patient must have a Wang Respiratory Score ≥ 5;
6. Patient who are hospitalized or in emergency/outpatient department and are expected to be hospitalized;
7. The parent/legal guardian must have provided written informed consent for the patient to participate.

Exclusion Criteria:

1. Patients who are less than 12 months old and whose head circumference is not within the normal range corresponding to their age and gender at the time of screening;
2. Patients who have received prohibited used drugs (except external preparations) specified in the protocol for a specified time.
3. Requires vasopressors or inotropic support at the time of enrollment;
4. Patients with known SARS-CoV-2 infection, influenza virus infection, mycoplasma infection or bacterial infection；
5. Patients with hypercapnia (Except for patients who have recovered at the time of screening);
6. Chronic or persistent feeding difficulties;
7. Concurrent gastrointestinal conditions that could seriously, in the opinion of the investigator, prejudice absorption of the Investigational Medicinal Product;
8. Symptomatic because of inborn errors of metabolism;
9. Bronchopulmonary dysplasia requiring assisted ventilationor with clinically significant congenital respiratory abnormalities, except for the result of RSV infection;
10. Patients with congenital heart disease (CHD) with significant hemodynamic changes, except simple CHD (such as patent ductus arteriosus, atrial septal defect or ventricular septal defect without hemodynamic influence).
11. Clinical evidence of hepatic decompensation
12. Renal failure including renal anomalies likely to be associated with renal insufficiency;
13. Patient is known to be HIV-positive (or the mother, if the potential patient is a child aged <6 months);
14. Suspected or known to have congenital acquired immunodeficiency;
15. A history of epilepsy or seizures;
16. A history of high allergies;
17. Any active or uncontrolled respiratory, cardiac, hepatic, central nervous system, or renal disease unrelated to RSV infection at baseline or any other medical condition that in the opinion of the investigator renders the patient unsuitable for enrollment;
18. Participation in an investigational drug or device study within 30 days prior to the date of screening;
19. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events during the study | From baseline through study completion, up to Day 26
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Subject withdrawals due to Adverse Events | From baseline through study completion, up to Day 26
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time to resolution of 6 clinical symptoms related to RSV infection | From baseline through study completion, up to Day 14
  Time to resolution of 6 clinical symptoms related to RSV infection
Time to resolution of individual clinical symptoms related to RSV infection | From baseline through study completion, up to Day 14
  Time to resolution of individual clinical symptoms related to RSV infection
Differences of the proportion of subjects with wheezing remission | From baseline up to Day2-7 and Day14
  Differences of the proportion of subjects with wheezing remission
Differences of the proportion of subjects with wheezing resolution | From baseline up to Day2-7 and Day14
  Differences of the proportion of subjects with wheezing resolution
Difference of the proportion of subjects with cough remission | From baseline up to Day2-7 and Day14
  Difference of the proportion of subjects with cough remission
Difference of the proportion of subjects with cough resolution | From baseline up to Day2-7、Day14 and D26
  Difference of the proportion of subjects with cough resolution
Changes of bronchiolitis score | From baseline up to Day2-7 and Day14
  The differences of change in the bronchiolitis score are to be evaluated between the Deuterium Hydrobromide for suspension and placebo arms after treatment. The total score is reported with a range from 0 to 12. The minimum and maximum values of 0 and 3 separately are defined for each scoring item. A decreasing value of the total score represents a clinical improvement. Subscales are not applicable in this scoring system.
Proportions of subjects achieving symptom remission &disease remission | From baseline up to Day2-7 and Day14
  Symptom remission was defined as bronchiolitis score ≤1. Disease remission was defined as bronchiolitis score ≤1 and with no assisted ventilation.
Time from first treatment to symptom remission &disease remission | From first treatment through study completion, up to Day 14
  The time difference from the first treatment to the time subjects achieved symptom remission between the Deuterium Hydrobromide for suspension and placebo arms.
  The time difference from the first treatment to the time subjects achieved disease remission between the Deuterium Hydrobromide for suspension and placebo arms.
Differences of frequency of Intensive Care Unit (ICU) admission | From first treatment through study completion, up to Day 14
  The differences of frequency of ICU admission between Deuterium Hydrobromide for suspension and placebo arms.
Differences of length of ICU stay | From first treatment through study completion, up to Day 14
  The differences of length of ICU stay between Deuterium Hydrobromide for suspension and placebo arms.
Differences of frequency of assisting ventilation | From first treatment through study completion, up to Day 14
  The frequency difference from the first treatment to the end of assisting ventilation therapy in subjects between the Deuterium Hydrobromide for suspension and placebo arms.
Differences in the duration of receiving oxygen therapy | From first treatment through study completion, up to Day 14
  The duration difference from the first treatment to the end of receiving oxygen therapy in subjects between the Deuterium Hydrobromide for suspension and placebo arms.
Changes of viral load | From baseline up to Day2-7 and Day14
  The antiviral effects in infants hospitalized with RSV are to be determined by measuring the differences in viral load determined by RT-PCR between the Deuterium Hydrobromide for suspension and placebo arms after treatment.
Changes of area under curve of viral load | From baseline up to Day2-7 and Day14
  The antiviral effects are to be determined by measuring the differences in area under curve (AUC).
Apparent total body clearance (CL/F) | From baseline up to Day2-7
  Apparent clearance of of 116-N1.
Area under the plasma concentration time curve from time zero to the last(AUC0-t) | From baseline up to Day2-7
  Area under the plasma concentration time curve from time zero to the last of 116-N1.
apparent volume of distribution(V) | From baseline up to Day2-7
  Apparent volume of distribution during the terminal phase of 116-N1.

SECONDARY OUTCOMES:
The correlation between viral load and the resolution time of 6 clinical signs related to RSV infection | From baseline up to Day2-7 and Day14
  Check if there is a positive correlation between viral load and the resolution time of 6 clinical signs
The correlation between viral load and bronchiolitis score | From baseline up to Day2-7and Day14
  Check if there is a positive correlation between changes in viral load and changes in bronchiolitis score.
The effect of the duration of RSV infection onset to the first use of the investigational drug on the treatment efficacy (clinical signs、change in bronchiolitis score from baseline) in subjects | From baseline up to Day2-7 and Day14
  The effect of the duration of RSV infection onset to the first use of the investigational drug on the treatment efficacy (clinical signs、change in bronchiolitis score from baseline) in subjects.
The difference in length of hospital stay | From baseline up to Day2-7 and Day14
  The difference in length of hospital stay between the experimental drug group and the placebo group due to RSV infection related diseases.
Proportions of subjects with viral load below LLOQ | From baseline up to Day2-7 and Day14
  The proportion of subjects whose viral load values are below LLOQ (lower limit of quantitation) after treatment.
The correlation between AUC0-t （ Area under the plasma concentration time curve from time zero to the last）and the resolution time of clinical signs | From baseline up to Day2-7 and Day14
  The correlation between AUC0-t （ Area under the plasma concentration time curve from time zero to the last）and the resolution time of clinical signs
The correlation between AUC0-t （ Area under the plasma concentration time curve from time zero to the last）and bronchiolitis score and RSV viral load (VL) in respiratory sample | From baseline up to Day2-7 and Day14
  The correlation between AUC0-t（ Area under the plasma concentration time curve from time zero to the last） and bronchiolitis score and RSV viral load (VL) in respiratory sample.

CONTACTS AND LOCATIONS:
Overall Officials: lanjuan li, Principal Investigator — Shulan (Hangzhou) Hospital; Zhen Qin, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (22):
- China (22):
  - The first Affiliated hospital of Bengbu Medical University, Bengbu, Anhui
  - Chongqing University Jiangjin Hospital, Chongqing, Chongqing Municipality
  - Xiamen Children's Hospital, Xiamen, Fujian
  - Xiamen Maternity and Child Healthcare Hospital, Xiamen, Fujian
  - Guangdong Women and Children's Hospital and Health Institute, Guangzhou, Guangdong
  - Panyu Maternal and Child care Service centre of Guangzhou, Guangzhou, Guangdong
  - The Sceond Affiliated hospital of Shantou University Medical college, Shantou, Guangdong
  - Shenzhen Guangming District People's Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Hainan women and children's Medical centre, Haikou, Hainan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Changde First people's Hospital, Changde, Hunan
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Maternal and Child Health, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linfen Central Hospital, Linfen, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Shulan (hangzhou) Hosipital, Hangzhou, Zhejiang
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou First people's Hospital, Hangzhou, Zhejiang